CLINICAL TRIAL: NCT00275093
Title: A Phase I Pharmacokinetic and Pharmacodynamic Study of Temsirolimus (CCI-779) in Patients With Advanced Malignancies and Normal and Impaired Liver Function: An NCI Organ Dysfunction Working Group Study
Brief Title: Temsirolimus in Treating Patients With Metastatic Solid Tumor or Lymphoma That Cannot Be Removed By Surgery Who Have Different Levels of Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03108; 04-04; U01CA069853 (NIH); U01CA062505 (NIH); U01CA099168 (NIH); U01CA062487 (NIH); U01CA062491 (NIH); U01CA062502 (NIH); CDR0000456257 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Hepatic Complications; Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Lymphoma | interventions — temsirolimus; Sirolimus

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of temsirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 12 patients are treated at the MTD.
  Interventions: Drug: temsirolimus; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of temsirolimus in treating patients with metastatic solid tumor or lymphoma that cannot be removed by surgery who have different levels of liver function. Temsirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Temsirolimus may have different effects in patients who have changes in their liver function

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety, tolerability, and to establish the maximum tolerated recommended dose (RD) CCI-779 (temsirolimus) in cohorts of patients with varying degrees of hepatic dysfunction (mild, moderate, and severe) in order to provide appropriate dosing recommendations for CCI-779 (temsirolimus) in this population.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetic (PK) profile of CCI-779 (temsirolimus) in patients with varying degrees of hepatic function.

II. To determine if the pharmacodynamic (PD) profile of CCI-779 (temsirolimus) as measured by drug effects on p70s6 kinase and p4EBP1 phosphorylation and other markers of mTOR inhibition in peripheral blood mononuclear cells (PBMC) is altered in patients with varying degrees of hepatic function.

III. To document the non-dose limiting toxicities and any anti-tumor efficacy associated with administration of CCI-779 (temsirolimus) in this patient population.

IV. To compare the NCI ODWG criteria and the Child-Pugh classification of hepatic dysfunction in terms of their predictive value in reducing interpatient variability in the PK and PD of CCI-779 (temsirolimus).

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to hepatic function (normal vs mild dysfunction vs moderate dysfunction vs severe dysfunction vs liver transplant).

Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of temsirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 12 patients are treated at the MTD.

After completion of study treatment, patients are followed periodically for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed solid tumor or lymphoma that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; all solid and lymphoma tumor types are eligible; patients with a liver mass (radiologically evident), elevated alpha-fetoprotein level (>= 500 ng/mL), and positive serology for viral hepatitis or history of alcoholic cirrhosis consistent with a diagnosis of hepatocellular carcinoma will be eligible without the need for pathologic confirmation of the diagnosis
* Life expectancy of >= 2 months
* ECOG performance status =< 2 (KPS >= 50)
* Absolute neutrophil count >= 1,000/mcl, and
* Platelets >= 100,000/mcl, and
* Serum creatinine =< 1.5 x ULN OR calculated creatinine clearance >= 60 mL/min/1.73 m^2
* Patients with abnormal liver function will be eligible and will be grouped according to total bilirubin and AST (SGOT); no distinction will be made between liver dysfunction due to metastases and liver dysfunction due to other causes; for patient stratification, liver function tests should be repeated within 72 hours of starting initial therapy
* Patients with biliary obstruction for which a shunt has been placed are eligible, provided the liver function tests have stabilized (two measurements at least tow days apart that put the patient in the same hepatic dysfunction stratum will be accepted as evidence of stable hepatic function); there must be no evidence of biliary sepsis and at least 2 weeks must have elapsed after the placement of a biliary shunt
* Patients receiving medications or substances with the potential to affect the activity the activity or pharmacokinetics of CCI-779 (temsirolimus), such as CYP3A4 substrates, inducers, or inhibitors may be enrolled at the discretion of the investigator; however, consideration should be given to stopping or switching to non-interfering agents if clinically feasible; in all cases, the use of these agents should be listed on the concomitant medication record
* The effects of CCI-779 (temsirolimus) on the developing human fetus and newborn are unknown; for this reason and because CCI-779 (temsirolimus) may be teratogenic, patients must not be pregnant or nursing; men or women of childbearing potential must have agreed to use an effective contraceptive method prior to study entry and for the duration of study participation; since interaction with CCI-779 (temsirolimus) and oral contraceptives is possible, a barrier method should be used and oral contraceptives are not permitted; a negative pregnancy test is required prior to starting therapy for women of childbearing age; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document in accordance with institutional and federal guidelines; all patients must be informed of the investigational nature of this study
* Patients must agree to undergo PK sampling and sample submission as outlined by the protocol

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, or immunotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from serious adverse events due to agents administered more than 4 weeks earlier
* Patients with a history of major surgery within 21 days prior to treatment
* Patients may not be receiving any other investigational agents
* Patients must not be planning to receive concurrent radiation, other chemotherapy, or immuno therapy for malignancy while receiving protocol treatment; hormonal treatment for prostate carcinoma may be continued and bisphosphonate treatment for bone disease is permitted
* Patients with unstable or untreated (non-irradiated) brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events; subjects with a prior history of CNS metastases will be eligible if the metastases have been treated with either RT or surgical resection ONLY and subjects are asymptomatic, with stable disease and no longer requiring steroids for at least 2 weeks; a screening magnetic resonance imaging (MRI)/CT (with contrast) is required
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to rapamycin or CCI-779 (temsirolimus)
* Uncontrolled serious intercurrent medical illness or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because CCI-779 (temsirolimus) is an agent with the potential for teratogenic or abortifacient effects; nursing women are also excluded, as there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CCI-779 (temsirolimus); breastfeeding should be discontinued if the mother is treated with CCI-779 (temsirolimus)
* HIV-positive patients receiving anti-retroviral therapy are excluded from the study due to the possibility of pharmacokinetic interactions with CCI-779 (temsirolimus); however, patients will not routinely be screened for HIV
* Patients who are currently receiving Rapamycin (RAP, Rapamune, Sirolimus) therapy are excluded from the study due to the possibility of overdosing, as CCI-779 is metabolized into sirolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-12; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
RD, defined as the highest dose level at which less than 33% of at least six patients experience DLT | 28 days

SECONDARY OUTCOMES:
PK profile of temsirolimus in patients with varying degrees of hepatic function | Days 1, 2, 4, 5, 8, 9, 11, 12, 15 of course 1
PD profile of temsirolimus as measured by drug effects on p70s6 kinase phosphorylation in PBMC | Days 1, 2, 4, and 8 course 1
Incidence of non-dose limiting toxicities | Up to 30 days
Antitumor efficacy | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: John Sarantopoulos, Principal Investigator — Cancer Therapy and Research Center at The UT Health Science Center at San Antonio
Locations (1):
- Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas, United States